CLINICAL TRIAL: NCT03233906
Title: Effects of Chia Seed Consumption on Body Composition, Blood Pressure, Blood Glucose, Satiety, Diet Displacement, Joint Pain, Mood and Serotonin Levels in Young, Healthy, Overweight/Obese Females
Brief Title: The Effects of Chia on Overweight/Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: California State Polytechnic University, Pomona (Other)
Responsible Party: Principal Investigator, Desiree Vera, Graduate Student, Human Nutrition and Food Science, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-16-188
Record Dates: First submitted 2017-07-17; First posted 2017-07-31 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Eating Behavior; Mood; Glucose; Dietary Modification
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Human subjects- females (18-45 y.o.) with a BMI greater than or equal to 26.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chia Seeds (Active Comparator): 10% of a participants total kcal estimated needs given in chia seeds everyday for 8 weeks.
  Interventions: Dietary Supplement: Chia Seeds- Salvia Hispanica
- Control (No Intervention): Habitual diet with avoidance of high fiber and high omega-3 fatty acid foods.

INTERVENTIONS:
Dietary Supplement: Chia Seeds- Salvia Hispanica — Chia seed added-10% of kcals and a no-chia control diet. 10% will be calculated using the following formula: Harris-Benedict equation multiplied by the activity factor of 1.2, 1.375, and 1.55 depending on each participant's activity level based on the information provided on the initial screening form.
  Arms: Chia Seeds

SUMMARY:
The purpose of the study is to examine the effect of chia seed consumption on body composition, blood pressure, blood glucose, satiety, mood, joint pain, and dietary displacement in overweight and obese females (18-45years). It is hypothesized that consuming chia seeds will bring about a positive change in body composition (lower % body fat), satiety, mood, joint pain, and blood pressure, lower blood glucose levels, increased fiber and improved nutrient intake, in overweight/ obese females.

DETAILED DESCRIPTION:
Specific Objectives: 1. Determine if chia seed diet addition of 10% of Kcals (CHIA) positively changes body composition in young, healthy, overweight/obese people (Tanita scale). A) Determine if CHIA will decrease blood pressure (monitor). 2. Determine if CHIA will decrease blood glucose (draw) 3. Determine if CHIA increases satiety and improves diet (recordings). 4. Determine if CHIA will decrease joint pain (questionnaire). 5. Determine if CHIA will increase positive mood changes (questionnaires) and increase blood serotonin levels (draw).

ELIGIBILITY:
Inclusion Criteria:

* are a female.
* are between the ages of 18 and 45.
* are not averse to consuming chia seeds on a regular basis (at least six weeks).
* have not taken any medication for any chronic disease (heart, diabetes, cancer) for twelve weeks.
* have not taken any steroid or hormone medication in the last eight weeks, excluding birth control pills...
* do not consume excess amounts of nuts and seeds. - do not consume alcohol on a regular basis.
* are not currently on a diet plan.
* are not pregnant or plan to become pregnant.

Exclusion Criteria:

* are a child, teenager, woman, or male younger than 18 or older than 45.
* eat large quantities of chia seeds on a regular basis.
* are taking any steroid or hormone medication (other than birth control pills). - are taking laxatives or fiber containing supplements on a regular basis.
* are pregnant or become pregnant.
* are currently on a diet plan.
* have a known allergy to seeds.
* consume excess amounts of seeds or nuts.
* consume alcohol on a regular basis.
* have a pacemaker or metal pins or plates in the body.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | baseline
  12-hour fasting plasma glucose levels will be assessed using a glucometer
Waist Circumference | baseline
  waist circumference will be measured for each participant
Caloric intake | baseline
  9, 3-day diet journals will be collected using a paper method
Serotonin | baseline
  Urine serotonin levels will be assessed
Body Weight | Baseline
  Tanita scale
Body Mass Index | Baseline
  Tanita sclae
Body Fat Percentage | Baseline
  Tanita scale
Fasting plasma glucose | week 4
  2-hour fasting plasma glucose levels will be assessed using a glucometer
Fasting plasma glucose | week 8
  2-hour fasting plasma glucose levels will be assessed using a glucometer
Waist Circumference | week 4
  waist circumference will be measured for each participant
Waist Circumference | week 8
  waist will be measured for each participant
Caloric intake | week 4
  9, 3-day diet journals will be collected using a paper method
Caloric intake | week 8
  9, 3-day diet journals will be collected using a paper method
Serotonin | week 4
  Urine serotonin levels will be assessed
Serotonin | week 8
  Urine serotonin levels will be assessed
Body Weight | week 4
  tanita scale
Body weight | week 8
  tanita scale
Body mass index | week 4
  tanita scale
body mass index | week 8
  tanita scale
Body fat percentage | week 4
  tanita scale
Body fat percentage | week 8
  tanita scale
Hip Circumference | Baseline
  Hip Circumference will be measured for each participant
Hip Circumference | week 4
  Hip Circumference will be measured for each participant
Hip Circumference | week 8
  Hip Circumference will be measured for each participant

SECONDARY OUTCOMES:
Blood Pressure | baseline
  Blood pressure will be taken using an automatic blood pressure machine
Blood Pressure | week 4
  Blood pressure will be taken using an automatic blood pressure machine
Blood Pressure | week 8
  Blood pressure will be taken using an automatic blood pressure machine
Joint Pain | baseline
  Joint pain will be assessed using The WOMAC (Western Ontario and McMaster Universities) Index of Osteoarthritis
Joint Pain | week 4
  Joint pain will be assessed using The WOMAC (Western Ontario and McMaster Universities) Index of Osteoarthritis
Joint Pain | week 8
  Joint pain will be assessed using The WOMAC (Western Ontario and McMaster Universities) Index of Osteoarthritis
Mood | Baseline
  Major Depression Inventory
Mood | week 4
  Major Depression Inventory
Mood | week 8
  Major Depression Inventory
Physical Activity | Baseline
  INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (August 2002) SHORT LAST 7 DAYS SELF-ADMINISTERED FORMAT
Physical Activity | week 4
  INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (August 2002) SHORT LAST 7 DAYS SELF-ADMINISTERED FORMAT
Physical Activity | week 8
  INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (August 2002) SHORT LAST 7 DAYS SELF-ADMINISTERED FORMAT
Sleep Quality | Baseline
  Measuring sleep quality using the Pittsburgh Sleep Quality Index
Sleep Quality | week 4
  Measuring sleep quality using the Pittsburgh Sleep Quality Index
Sleep Quality | week 8
  Measuring sleep quality using the Pittsburgh Sleep Quality Index
Fat mass | Baseline
  using a tanita scale
Fat mass | week 4
  using a tanita scale
Fat mass | week 8
  using a tanita scale
Fat Free Mass | Baseline
  using a tanita scale
Fat Free Mass | week 4
  using a tanita scale
Fat Free Mass | week 8
  using a tanita scale
Total body water | Baseline
  using a tanita scale
Total body water | week 4
  using a tanita scale
Total body water | week 8
  using a tanita scale
Macro nutrient intake | Baseline
  3, 3-day diet journals will be collected using a paper method
Macro nutrient intake | week 4
  3, 3-day diet journals will be collected using a paper method
Macro nutrient intake | week 8
  3, 3-day diet journals will be collected using a paper method
Micronutrient intake | Baseline
  3, 3-day diet journals will be collected using a paper method
Micronutrient intake | week 4
  3, 3-day diet journals will be collected using a paper method
Micronutrient intake | week 8
  3, 3-day diet journals will be collected using a paper method
Dietary intake Satiety | Baseline
  3, 3-day diet journals will be collected using a paper method
Dietary intake Satiety | week 4
  3, 3-day diet journals will be collected using a paper method
Dietary intake Satiety | week 8
  3, 3-day diet journals will be collected using a paper method
Dietary intake displacement | Baseline
  3, 3-day diet journals will be collected using a paper method
Dietary intake displacement | week 4
  3, 3-day diet journals will be collected using a paper method
Dietary intake displacement | week 8
  3, 3-day diet journals will be collected using a paper method

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Burns-Whitmore, DrPh, RD, Study Director — California State Polytechnic University, Pomona
Locations (1):
- California State Polytechnic University, Pomona, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No